CLINICAL TRIAL: NCT02299752
Title: Double Gloves: A Randomized Trial to Evaluate a Simple Strategy to Reduce Contamination During Resuscitation
Brief Title: Unnoticed Gloves Perforation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gloves/2014/01
Record Dates: First submitted 2014-11-13; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Catheterization; Contamination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Catheterization (Experimental): Blood vessel Catheterization during resuscitation with single and double - gloving system. Catheterization was performed using simulation mannikin
  Interventions: Procedure: single-gloving system; Procedure: double-gloving system

INTERVENTIONS:
Procedure: single-gloving system — single-gloving system was used during Catheterization
Procedure: double-gloving system — double-gloving system was used during Catheterization. inner and outer gloves were the same size

SUMMARY:
The aim of the study was to investigate the incidence of glove perforation in cannulation of blood vessels (CBV) during resuscitation and compare perforation rates between single and double-gloves.

DETAILED DESCRIPTION:
Exposure to blood pathogens among medical staff is a serious problem that should be first and foremost prevented . The risk of acquiring a virus from one percutaneous needle stick is 0.3% to 0.4% for human immunodeficiency virus (HIV), 6% to 30% for hepatitis B (HBV), and 2.7% to 10% for hepatitis C (HCV). The prevention of blood-borne infections is particularly important during cases when emergency medical attention is needed. Emergency Response Personnel that work in this profession have taken medical rescue courses to prepare for situations of sudden health threats, hence the majority of procedures is associated with direct contact with body fluids of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* Medical profession (paramedics, nurses, physicians) or medical students (nurses, paramedics, physicians)

Exclusion Criteria:

* Not meet the above criteria
* Wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
visible puncture | 1 day
  Checking gloves for visible damage in the course of cannulation during resuscitation

SECONDARY OUTCOMES:
WLT | 1 day
  Water leak test was used to checking unnoticed gloves damage

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland